CLINICAL TRIAL: NCT00639002
Title: A Phase 2, Two Stage, Open-label, Clinical Trial to Determine the Therapeutic Effect and Safety of an Oral JAK2-inhibitor (INCB018424) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study to Determine the Effect and Safety of an Oral Janus Kinase 2 (JAK2)-Inhibitor (Ruxolitinib; INBC018424) in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-255
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ruxolitinib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib then Ruxolitinib + Dexamethasone (Experimental): Patients received ruxolitinib 25 mg orally twice daily (bid) in each treatment cycle of 28 days. For those patients who had disease progression at any time or stable disease for 3 cycles and did not meet a withdrawal criterion, or withdrew consent, then 40 mg of dexamethasone was added to ruxolitinib on Days 1 to 4, 9 to 12, and 17 to 20 of four 28-day cycles. After the 4th cycle, 40 mg of dexamethasone was administered only on Days 1 to 4 of each subsequent cycle. Patients could continue to receive monotherapy or combination therapy indefinitely as long as no withdrawal criterion was met, did not have progressive disease and were receiving some clinical benefit.
  Interventions: Drug: Ruxolitinib 25 mg; Drug: Dexamethasone 40 mg

INTERVENTIONS:
Drug: Ruxolitinib 25 mg — Ruxolitinib was supplied as 5 and 25 mg tablets.
  Other Names: INCB018424
Drug: Dexamethasone 40 mg — Dexamethasone was obtained commercially by Investigators in tablet strengths of 20 or 40 mg.

SUMMARY:
The purpose of this study was to determine clinical efficacy and safety of ruxolitinib (INCB018424), a small molecule Janus kinase 2 (JAK2)-inhibitor, in patients with refractory or relapsed multiple myeloma.

DETAILED DESCRIPTION:
The protocol was originally designed as a Simon two stage but after it was determined that the initial 13 patients enrolled did not meet the definition of a 'responder' according to the International Uniform Response Criteria for multiple myeloma the protocol was amended to allow patients who had disease progression at any time or stable disease for 3 cycles and did not meet a withdrawal criterion or had withdrawn consent to have 40 mg of dexamethasone added to their dose of ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma with evidence of measurable disease.
* Relapsed or refractory disease with at least one line of prior therapy.
* Adequate bone marrow reserve.

Exclusion Criteria:

* Received anti-cancer medications or investigational therapy in the past 28 days.
* Intracranial disease or epidural disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Jagannath, MD, Principal Investigator — St. Vincent's Comprehensive Cancer Center, New York, New York
Locations (3):
- United States (3):
  - Highland, California
  - Boynton Beach, Florida
  - New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruxolitinib Then Ruxolitinib + Dexamethasone: Patients received ruxolitinib 25 mg orally twice daily (bid) in each treatment cycle of 28 days. For those patients who had disease progression at any time or stable disease for 3 cycles and did not meet a withdrawal criterion or withdrew consent then 40 mg of dexamethasone was added to ruxolitinib on Days 1 to 4, 9 to 12, and 17 to 20 for four 28-day cycles. After the 4th cycle, 40 mg of dexamethasone was administered only on Days 1 to 4 of each subsequent cycle. Patients could continue to receive monotherapy or combination therapy indefinitely as long as no withdrawal criterion was met, did not have progressive disease and were receiving some clinical benefit.
Period: Overall Study
Arm/Group | Ruxolitinib Then Ruxolitinib + Dexamethasone
Started | 13
Received Ruxolitinib | 13
Received Ruxolitinib + Dexamethasone | 7
Completed | 0
Not Completed | 13
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Disease progression | 3
Not completed — Physician Decision | 6
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib Then Ruxolitinib + Dexamethasone
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Stage I: Relatively few cancer cells have spread throughout the body. Levels of red blood cells and calcium in the blood are normal. No bone tumors. M-protein in the blood or urine is very low. Possibly no symptoms of disease.
  Stage II: A moderate number of cancer cells have spread throughout the body.
  Stage III: A large number of cancer cells have spread throughout the body. There may be 1 or more of the following:
  * Decreased red blood cells, causing anemia
  * High amounts of calcium in the blood
  * More than 3 bone tumors (plasmacytomas)
  * High levels of M-protein in blood or urine
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 10
    More than one race | 0
    Unknown or Not Reported | 0
Stage of multiple myeloma at initial diagnosis [Number; unit: participants]
  I | 0
  II | 4
  III | 4
  Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders According to the International Uniform Response Criteria for Multiple Myeloma
Description: A responder is defined as a patient with a complete response (negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow) or a partial response (≥ 50% reduction of serum M-protein and reduction in 24 h urinary M-protein by ≥ 90% or to < 200 mg per 24 h).
Time Frame: Day 1 of Cycles 2, 3, and 4 and then every 3 months thereafter (up to 25 months).
Population: Intent-to-treat population: All patients who were enrolled and took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Ruxolitinib Then Ruxolitinib + Dexamethasone
Number analyzed (Participants) | 13
participants | 0

2. Secondary Outcome: Time to Disease Progression According to the International Uniform Response Criteria for Multiple Myeloma
Description: Progressive Disease requires 1 or more of the following:
  Increase of ≥ 25% from baseline in:
  Serum M-component and/or (increase ≥ 0.5 g/dL).
  Urine M-component and/or (increase ≥ 200 mg/24 h).
  In patients without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels increase must be > l0 mg/dL.
  Bone marrow plasma cell percentage ≥ 10%.
  Definite development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas.
  Development of hypercalcemia.
Time Frame: Day 1 of Cycles 2, 3, and 4 and then every 3 months thereafter (up to 25 months).
Population: Intent-to-treat population. This outcome measure was not analyzed as no patients achieved a response.
Arm/Group | Ruxolitinib Then Ruxolitinib + Dexamethasone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to end of study
Description: Safety population: All subjects who were enrolled and took at least 1 dose of study medication.
Groups:
- Ruxolitinib: Patients received ruxolitinib 25 mg orally twice daily (bid) in each treatment cycle of 28 days until the following criteria were met: Disease progression at any time or stable disease for 3 cycles and did not meet a withdrawal criterion, or withdrew consent.
- Ruxolitinib + Dexamethasone: Following administration of ruxolitinib 25 mg bid alone, for those patients who had disease progression at any time, stable disease for 3 cycles, did not meet a withdrawal criterion, or withdrew consent, then 40 mg of dexamethasone was added to ruxolitinib on Days 1 to 4, 9 to 12, and 17 to 20 of four 28-day cycles. After the 4th cycle, 40 mg of dexamethasone was administered only on Days 1 to 4 of each subsequent cycle. Patients could continue to receive monotherapy or combination therapy indefinitely as long as no withdrawal criterion was met, did not have progressive disease and were receiving some clinical benefit.
Arm/Group | Ruxolitinib | Ruxolitinib + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 6/13 | 6/7
Other Adverse Events (participants affected / at risk) | 11/13 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=13) | Ruxolitinib + Dexamethasone (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Disease progression (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=13) | Ruxolitinib + Dexamethasone (N=7)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Entropion (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 4 | 2
Pyrexia (General disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Oral infection (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Candidiasis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Blood creatinine increased (Investigations) | 4 | 2
Haemoglobin decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood calcium increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1
Breath sounds abnormal (Investigations) | 0 | 1
Sputum culture positive (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.